CLINICAL TRIAL: NCT02181374
Title: The Diagnosis Value of Serum Marker in Stroke Associated With Nonvalvular Atrial Fibrillation
Acronym: CE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Xijing-25
Record Dates: First submitted 2014-06-03; First posted 2014-07-03 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Ischemic Stroke
Keywords: atrial fibrillation; NT-proBNP; Cardioembolic Stroke
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Embolic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — NT-proBNP
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the diagnostic value of serum NT - proBNP in stroke associated with nonvalvular atrial fibrilltion.

DETAILED DESCRIPTION:
All included in the cases in 7 days of blood samples, the detection of serum NT - proBNP.Through the single factor analysis to determine the serum NT - proBNP central source sex stroke prediction values.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ Age ≤ 85;
* Meet the clinical diagnostic criteria for acute ischemic stroke;
* onset within 7 days;

Exclusion Criteria:

* Severe systemic disease (chronic inflammation, infection, blood system diseases, cancer, kidney failure, liver failure,heart failure);
* Nearly a month history of myocardial infarction;
* pregnant;
* Serious neurological disease that the diagnosis is unclear;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 ≤ Age ≤ 85; meet the clinical diagnostic criteria for acute ischemic stroke; onset within 24 hours at the same time more than one hour; it was diagnosed with experiential doctor.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value of serum NT - proBNP in stroke associated with nonvalvular atrial fibrilltion | 34 months
  All included in the cases in 7 days of blood samples , the detection of serum NT - proBNP.Through the single factor analysis to determine the prediction values of serum NT - proBNP in stroke associated with nonvalvular atrial fibrilltion.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, MD, Study Director — The Department of Neurology, Xijing Hospital
Locations (1):
- The Department of Neurology, Xijing Hospital, Xi'an, Shaanxi, China